CLINICAL TRIAL: NCT05789849
Title: Data Collection for Validation of a Noninvasive Blood Pressure Auscultatory Algorithm - Pregnant Women
Brief Title: Data Collection for Validation of an NIBP Algorithm in Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 219397851
Record Dates: First submitted 2023-03-16; First posted 2023-03-29 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Blood Pressure

STUDY DESIGN:
Intervention Model Description: This is an open label, single-site, single arm, prospective, pivotal study including a training phase and a data collection phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Blood Pressure Collection (Experimental): This study has only 1 arm; investigational NIBP measurements will be collected using a NIBP Auscultatory Algorithm with alternating NIBP measurements collected using a reference sphygmomanometer.
  Interventions: Device: Collecting blood pressure measurements with noninvasive blood pressure device

INTERVENTIONS:
Device: Collecting blood pressure measurements with noninvasive blood pressure device — Noninvasive blood pressure measurements will collected based on the recommendations of the International Organization for Standardization (ISO) 81060-2:2018+A1:2020 Non-invasive sphygmomanometers -Clinical investigation of intermittent automated measurement type. This study has only 1 arm; investigational NIBP measurements will be collected using a NIBP Auscultatory Algorithm with alternating NIBP measurements collected using a reference sphygmomanometer.
  Other Names: GE DINAMAP® SuperSTAT algorithm

SUMMARY:
The purpose of the study is to collect per subject blood pressure data on the device's intended population as described in the International Organization for Standardization (ISO) Standard 81060-2:2018+A1:2020 Non-invasive sphygmomanometers.

DETAILED DESCRIPTION:
The purpose of the study is to collect data per subject NIBP measurements by (1) oscillometric means using the GE NIBP Auscultatory Algorithm and (2) by conventional auscultatory means in a pregnant population. These measurements include Systolic BP (mmHg) and Diastolic BP (mmHg). The secondary objective of this study is to collect per procedure and log files from the device. The safety objective of this study is to collect safety information, including type and number of adverse events, serious adverse events and device issues.

This is an open label, single-site, single arm, prospective, pivotal study including a training phase and a validation phase with demographics-based stratification quota. Subjects are sequentially tested with investigational and reference blood pressure measurements.

ELIGIBILITY:
Inclusion Criteria:

Are pregnant female volunteers aged 18 years or older;

Gestation beyond the first trimester as evidenced by gestational age of greater than or equal to 14 weeks and 0 days;

Have compatible anatomy to fit a standard air-filled occlusive cuff size (an upper limb circumference ranging 17 cm to 40 cm);

Are willing and able to volunteer to provide multiple blood pressure measurements as required for study procedures;

Are able and willing to provide written informed consent.

Exclusion Criteria:

Exhibit signs or symptoms or have a current diagnosis of peripheral vascular disease;

Have current, uncontrolled circulatory shock or cardiac arrhythmias that pose risk to the patient or could interfere with completion of study blood pressure determinations;

Exhibit injuries, deformities, intravenous lines, or other abnormalities that, in the opinion of the investigator, may prevent proper occlusive cuff application or functioning; the investigator, may prevent proper occlusive cuff application or functioning;

Have contraindications to blood pressure measurement methods used in the study or any medical condition where study procedures could pose a risk to the subject/patient's physiological stability, in the opinion of a medically qualified investigator.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Collection of per subject NIBP measurements | Start of blood pressure acquisition until three valid pairs obtained, approximately one hour
  The primary objective of this study is to collect per subject NIBP measurements by oscillometric means using the GE NIBP Auscultatory Algorithm and by conventional auscultatory means in a pregnant population. These measurements include both Systolic BP (mmHg) and Diastolic BP (mmHg).

SECONDARY OUTCOMES:
Collection of per procedure and device log files. | Start of blood pressure acquisition until three valid pairs obtained, approximately one hour
  The secondary objective of this study is to collect per procedure and device log files.

OTHER OUTCOMES:
Number of Safety Events and Device Issues | Start of blood pressure acquisition until three valid pairs obtained, approximately one hour
  The safety objective of this study is to collect safety information, including type and number of adverse events, serious adverse events, and device issues.

CONTACTS AND LOCATIONS:
Overall Officials: Nandini Raghuraman, MD, Principal Investigator — Division of Maternal-Fetal Medicine Washington University in St Louis School of Medicine; Adithya Bhat, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No